CLINICAL TRIAL: NCT04254627
Title: Tumor Necrosis Factor (TNF) and Glucocorticoid Antagonist for Gulf War Illness (GWI)-Associated Multi-symptom Disease Homeostasis Reset
Brief Title: TNF and Glucocorticoid Antagonist for GWI Associated Multi-symptom Disease Homeostasis Reset
Acronym: E/M
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: RTI International (Other); Miami VA Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GWICTIC-EMphase1; CDMRP-PC16GW170044 (Other Grant/Funding Number: U.S. Army Medical Research and Materiel Command)
Record Dates: First submitted 2020-01-09; First posted 2020-02-05 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Gulf War Illness
Keywords: Gulf War Illness; Veterans; etanercept; mifepristone; VA Healthcare; TNF; Multi-symptom disease; Phase I
MeSH Terms: interventions — Etanercept; Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mifepristone 300 mg (Experimental): All participants will receive etanercept 50 mg weekly for 12 weeks. After completion of the etanercept course, participants will be randomized between two Arms of mifepristone. Participants randomized to Arm 1 will receive one week of mifepristone at 300 mg daily.
  Interventions: Drug: Etanercept; Drug: Mifepristone
- Mifepristone 600 mg (Experimental): All participants will receive etanercept 50 mg weekly for 12 weeks. After completion of the etanercept course, participants will be randomized between two Arms of mifepristone. Participants randomized to Arm 2 will receive one week of mifepristone at 600 mg (2x300 mg) daily.
  Interventions: Drug: Etanercept; Drug: Mifepristone

INTERVENTIONS:
Drug: Etanercept — Etanercept 50 mg weekly injection
  Other Names: Enbrel
Drug: Mifepristone — Mifepristone 300 mg pill
  Other Names: Mifeprex; RU-486

SUMMARY:
Gulf War Illness is a condition that affects multiple major organ systems, resulting in a diverse array of symptoms that include debilitating fatigue, memory and cognition difficulties, headaches, sleep disturbances, gastrointestinal problems, skin rashes, and musculoskeletal/joint pain. This phase I single-site, open-label two-arm study will assess the safety and mechanistic efficacy of a sequential etanercept-mifepristone intervention for Gulf War Illness. The results of this phase I study will be compared to those from an existing short-duration study to identify the optimal duration and dosage for use in a future phase II study.

DETAILED DESCRIPTION:
This is a study in male Veterans 45-70 years of age who meet the modified Kansas and Centers for Disease Control and Prevention (CDC) criteria for GWI (Gulf War Illness) and have high physiologic stress. This phase I single-site, open-label, two-arm study will focus on optimizing the dosage of a sequential etanercept-mifepristone intervention for GWI. Twenty participants will be assessed at baseline, 6, 12, 13, 16 and 24 weeks. The investigators will use systems biology methods to perform computational modelling of physiological responses to supervised maximal exercise challenge studies on a fitness bicycle at baseline and 24 weeks. These analyses will assess the impact of the treatment on homeostatic networks: the changes in levels of physiological parameters and the changes in inter-correlations among the measured parameters (e.g., cytokines), cross-sectionally and over time. Participants will also undergo subjective assessments of functional health, symptom severity, pain, fatigue, and cognition at baseline, 6, 12, 13, 16, and 24 weeks. Participants will be observed through the treatment period and for 3 months after completion to assess immediate effects and durability of the response.

The results of this phase I study will be compared to those from an existing short-duration study to identify the optimal duration and dosage for use in a future phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. 45-70 years old,
2. Male sex,
3. In good health by medical history prior to 1990
4. Meets modified Kansas and CDC case definition criteria for Gulf War Illness. Original Kansas criteria and CDC case definitions, including their exclusionary conditions. The modified Kansas definition, which includes the CDC criteria, includes the following:

   1. Fatigue after exercise as predominant component (a history of exercise intolerance or exercise-induced worsening of symptoms)
   2. Allowance for normal illnesses of aging, such as hypertension and diabetes, if the conditions are treated and are in demonstrable stable and normal ranges at the time of screening and assessment.
   3. Allowance of stable comorbid conditions such as PTSD, MDD, and TBI that have not required hospitalization in the 5 years prior to recruitment. Severe TBI is excluded.
5. Able to provide consent to study,
6. Subjects of childbearing potential must practice effective contraception during the study, and be willing to continue contraception for at least 6 months after intervention.
7. Agrees to participate in follow-up visits.

Exclusion Criteria:

1. Current treated or untreated major depression with psychotic or melancholic features, schizophrenia, bipolar disorder, delusional disorders, dementias of any type, and alcoholism or drug abuse (as determined by self-report, SAGE-SR, and Ham-D)
2. Known allergy to mifepristone, misoprostol, or medicines that contain misoprostol, such as Cytotec or Arthrotec.
3. Current heavy alcohol or tobacco use (self-report). Alcohol consumption not to exceed approximately 15 drinks per week (with a drink defined as 12 oz beer, 5 oz wine, or 1.5 oz distilled spirits) and tobacco use not to exceed 20 cigarettes (or equivalent) per day.
4. Current organ failure (as determined by metabolic panel and self-report)
5. Current treated or untreated rheumatologic and inflammatory disorders, as determined by medical diagnosis of one or more of the following: osteoarthritis, rheumatoid arthritis (RA), lupus, spondyloarthropathies -- ankylosing spondylitis (AS) and psoriatic arthritis (PsA), Sjogren's syndrome, gout, scleroderma, infectious arthritis, and polymyalgia rheumatic
6. Chronic active infections such as HIV, hepatitis B, and hepatitis C (as determined by antibody tests
7. History of organ transplant (self-report)
8. Current untreated primary sleep disorders such as insomnias, sleep related breathing disorders, etc. (self-report)
9. History of tuberculosis exposure (determined by QuantiFERON-TB® positivity)
10. Use of medications that could affect immune function (e.g., steroids, immunosuppressants) or limit the interpretation of the exercise challenge (self- report)
11. Renal disease (self-report; laboratory results: renal insufficiency with serum creatinine > 2.0 mg/dL or eGFR < 44; or currently on renal dialysis).
12. Hepatic insufficiency (bilirubin >2.5mg/dL or transaminases >5x the ULN) Subjects with Gilberts syndrome are eligible for the study if other liver function tests are normal, regardless of bilirubin level.
13. Currently have no exclusionary diagnoses that could reasonably explain the symptoms of their fatiguing illness and their severity, using the exclusion criteria best described in the Ambiguities in case definition paper for Chronic Fatigue Syndrome (CFS) which clarifies exclusionary conditions.
14. Are scheduled for surgery within 24 weeks of study enrollment.
15. Cushing's disease or salivary cortisol level greater than 0.812 ug/dL.
16. QT prolongation, as evidenced by medical history (self-report) or ECG at screening.
17. Uncontrolled diabetes (A1c>7.5).

Prohibited concomitant or prior therapies:

1. Immunosuppressant drugs, including glucocorticoid taper, topical/inhaled glucocorticoids
2. Currently on dialysis
3. Recipient of bone marrow or organ transplant
4. Previous or current treatment with angiogenic growth factors, cytokines, gene or stem cell therapy
5. Participating in another interventional clinical trial of an investigational therapy within 8 weeks prior to consent to participate in this study, or planning to participate in another interventional clinical trial of an investigational therapy within 26 weeks after consent to participate in this study
6. Any herbal medicine that contains licorice root.
7. Selective Blood thinners:

   * Only Apixaban and Warfarin will be included. Rivaroxaban cannot be included as there are higher drug to drug interactions as well as Apixaban 2.5 mg BID.
   * If a participant is on Warfarin, a baseline INR will be obtained, the Warfarin dose will be reduced and an INR will be rechecked 48-72 hours after starting Mifepristone.
   * If a participant is on Apixaban, the dose must be reduced by 50%.
   * Please note that if participants are taking anticoagulants, there is a potential interaction that could lead to possible increased on risk of bleeding and will require more frequent monitoring by the Coordinator.

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Safety - incidence and severity of adverse events | 16 weeks
  Safety is assessed by the incidence and severity of adverse events, by relation to the study intervention.
Mechanistic effects on biomarker relationships | Baseline and 24 weeks
  Mechanistic effects on biomarker network dynamics are measured by the change in median summary score for network-level distance between the Gulf War Illness biomarker profile at rest and model-predicted stable (healthy) states. These summary scores have a minimum value of zero and reflect the overall difference between the multidimensional relationships of the immune, autonomic, and neuroendocrine systems of ill participants at rest, relative to predicted values for stable (healthy) states. The analysis will be completed using the results of physical measures and biomarker assays performed on blood draws taken at rest prior to exercise challenges at baseline and 16 weeks. These include a Gulf War Illness-specific nanostring gene expression platform, an 18-multiplex cytokine assay, flow cytometry, neuropeptide, sex and stress hormone panels, and physical autonomic measures. Decreases in summary scores between baseline and 24 weeks indicate a better outcome.

SECONDARY OUTCOMES:
Homeostatic network correction | Baseline and 24 weeks
  The degree of correction of the homeostatic network toward normal is measured by the median summary score for network-level differences in connectivity of biomarker networks at multiple times during dynamic exercise challenges. These summary scores have a minimum value of zero and reflect overall changes within the immune, autonomic, and neuroendocrine systems during exercise, relative to predicted values for stable (healthy) states. The analysis will use the results of physical measures and blood draws taken before, during, and after exercise challenges at baseline and 24 weeks. The biomarker assays and physical measures include a Gulf War Illness-specific nanostring gene expression platform, an 18-multiplex cytokine assay, flow cytometry, neuropeptide, sex and stress hormone panels, and physical autonomic measures at multiple times during each exercise challenge and 24 hours afterward. Decreases in summary scores between baseline and 16 weeks indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Klimas, MD, Principal Investigator — Miami VA Healthcare System
Locations (2):
- United States (2):
  - Nova Southeastern University, Davie, Florida
  - Miami VA Healthcare System, Miami, Florida

IPD SHARING:
Plan to Share IPD: No
The plan is to release primary results from the study to ClinicalTrials.gov. Data are the property of Nova Southeastern University, but data and publication thereof will not be unduly withheld. Those interested in E/M data should reach out to Nancy Klimas (PI) for more information.